CLINICAL TRIAL: NCT01277133
Title: The Correlation Between the Moment of Bevacizumab theRapy initiatiOn and the Efficacy in patieNt With Metastatic Breast Cancer Treated With First Line Regimens Based On AvaStin
Brief Title: An Observational Study on The Correlation Between Time of Initiation of Avastin (Bevacizumab) Treatment And Progression-Free Survival in Patients With Metastatic Breast Cancer (CRONOS 2)
Status: Terminated | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25191
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This single arm, prospective, observational study will assess the correlation between the time from start of chemotherapy to the start of Avastin (bevacizumab) treatment with progression-free survival in patients with previously untreated metastatic breast cancer. Patients will be followed for up to 12 months after progressive disease occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Previously untreated metastatic breast cancer
* Scheduled to start 1st line chemotherapeutic treatment
* ECOG performance status 0-1

Exclusion Criteria:

* Any conditions included in contraindication list for Avastin
* Prior chemotherapy for metastatic breast cancer
* Adjuvant/neoadjuvant chemotherapy or radio-chemotherapy of non-metastatic malignancy completed <6 months prior to treatment start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with metastatic HER2 negative breast cancer. First-line treatment with Avastin
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2010-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Correlation between the time from start of chemotherapy to the start of Avastin treatment with progression-free survival | 60 months

SECONDARY OUTCOMES:
Overall survival | 60 months
Safety: Incidence of adverse events | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Cluj-Napoca, Romania